CLINICAL TRIAL: NCT06529432
Title: Efficacy, Safety and Pharmacokinetics of Bupivacaine Liposome Injection for Paravertebral Nerve Block in the Treatment of Postoperative Pain After Thoracoscopic Surgery: a Multicenter, Randomized, Double-blind, Dose-finding, Positive Control, Phase Ⅱ Clinical Trial
Brief Title: A Study of Bupivacaine Liposome Injection in the Treatment of Pain After Thoracoscopic Surgery
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BULI-201
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Local Analgesia Via Nerve Block
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: A multicenter, randomized, double-blind, dose-finding, positive control, phase Ⅱ clinical trial of liposomal bupivacaine injection
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine Liposome Injection (Experimental)
  Interventions: Drug: Bupivacaine Liposome Injection
- Bupivacaine Hydrochloride Injection (Active Comparator)
  Interventions: Drug: Bupivacaine Hydrochloride Injection

INTERVENTIONS:
Drug: Bupivacaine Liposome Injection — Bupivacaine Liposome Injection Low Dose or Moderate Dose or High Dose
  Arms: Bupivacaine Liposome Injection
Drug: Bupivacaine Hydrochloride Injection — Bupivacaine Hydrochloride Injection Low Dose or Moderate Dose or High Dose
  Arms: Bupivacaine Hydrochloride Injection

SUMMARY:
The objective of this study is to evaluate the efficacy, safety, and tolerability of bupivacaine liposomes for paravertebral nerve block in the treatment of thoracoscopic postoperative pain, and to evaluate the relevant human pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

-

1. Subjects who are willing to strictly follow the clinical trial protocol to complete this study and voluntarily sign informed consent;
2. Elective surgical subjects undergoing lobectomy by single-aperture thoracoscope under general anesthesia;
3. age ≥18 years old , Male or female.
4. 18 kg/m2≤BMI≤30 kg/m2.
5. ASA Physical Status Classification I-II.

   Exclusion Criteria:

   - Participants with any of the following criteria were excluded from the study：

1. Pre-existing and combined diseases:

1. Subjects with a history of myocardial infarction or unstable angina pectoris, or a history of severe arrhythmias such as atrioventricular block of degree II and above, or NYHA grade II and above in the 6 months before randomization.
2. Subjects with a history of ischemic stroke or transient ischemic attack (TIA).
3. Subjects with psychiatric disorders (such as schizophrenia, depression, etc.) and cognitive dysfunction.
4. Subjects with sensory disorders such as hyperalgesia.
5. Subjects with other physical pain witch may affect the evaluation of postoperative pain.
6. Subjects with airway or spinal anatomic factors caused by obstruction of ventilation, bronchiectasis, severe intraoperative thoracic adhesion, etc.

2. Laboratory and other tests:

1. Abnormal laboratory results during screening. • Fasting blood glucose (FPG) ≥10.0mmol/L.

   • Abnormal liver function: aspartate aminotransferase (AST) or/and alanine aminotransferase (ALT) and/or total bilirubin (TBIL) ≥1.5×ULN.

   • Abnormal renal function: serum creatinine (Cr) ≥1.5×ULN, or dialysis subjects.

   • Abnormal coagulation function: PT> upper normal value +3s and/or APTT > upper normal value +10s.

   • Platelet (PLT) <80×109/L.

   • Hemoglobin concentration (Hb) < 70g/L.
2. Screening period heart rate < 50 beats/min or heart rate > 100 beats/min; 12-lead ECG QTc interval prolonged: male ≥450ms, female ≥470ms.
3. Subjects with refractory hypertension or a history of refractory hypertension before randomization.

3. Combined drugs:

(1) Subjects who allergic to or contraindicated with bupivacaine, other amide local anesthetics, and other drugs that may be used during the trial (e.g., propofol, remazolam, opioids, etc.).

(2) Subjects who used any of the following drugs within 5 drug half-lives prior before randomization (drug half-lives are based on actual drug instructions, or at least 48 hours of elution if half-lives are unknown):

* Class III antiarrhythmic drugs such as amiodarone.
* Drugs that affect liver metabolism: strong CYP1A2 inhibitors such as ciprofloxacin, enoxacin, fluvoxamine; CYP1A2 substrates: such as theophylline, imipramine; Strong CYP3A4 inhibitors such as voriconazole, ketoconazole, Ritonavir; CYP3A4 substrates such as darunavir, Indinavir, saquinavir; Strong CYP3A4 inducers such as rifampin.
* Intravenous or oral corticosteroids.
* Sedative drugs: benzodiazepines (such as diazepam, flurazepam, oxazepam, cloazepine, triazolam, alprazolam, esazolam, midazolam, etc.), barbiturates, carbamazepine, phenytoin, magnesium sulfate, chloral hydrate, etc..
* Pain relief and other drugs: Nonsteroidal anti-inflammatory drugs (aspirin is permitted for the prevention of cardiovascular events, provided it is used steadily for at least 30 days prior to randomization, Daily dose ≤100mg/ day), opioid agonists/antagonists, central alpha-adrenergic agonists (e.g. Clonidine, dexmedetomidine), anticonvulsants (e.g. Carbamazepine, pregabalin, gabapentin), antidepressants (e.g. Tricyclic, selective 5-HT reuptake inhibitors).

  4. Others:
  1. Subjects had a history of substance abuse, drug use, and/or alcohol abuse within the 1 year prior to randomization, with alcohol abuse defined as drinking an average of more than 2 units of alcohol per day (1 unit =360mL beer or 45mL liquor with 40% alcohol or 150 ml wine); Or consume alcoholic food or drink within 24 hours before receiving the study drug.
  2. Subjects consumed excessive amounts of tea, coffee, grapefruit/grapefruit juice, grapefruit juice, caffeinated beverages (averaging more than 8 cups per day, 200 mL per cup) in the 14 days prior to randomization.
  3. Female subjects who are pregnant or breastfeeding.
  4. Subjects who have planned to have children within 30 days prior to the screening period and have planned to have children within six months from the date of signing the informed consent to the last use of the investigational drug and are unwilling or unable to use effective contraception.
  5. Subjects who have participated in other clinical trials as subjects, and/or previously received investigational drug or device in this clinical trial within the 3 months prior to randomization.
  6. Subjects who have any other factors deemed unsuitable for participation in this trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-08-21 (Estimated); Primary Completion 2026-09-28 (Estimated); Study Completion 2026-10-12 (Estimated)

PRIMARY OUTCOMES:
Area under the time curve of pain intensity during exercise (or cough) for 72 hours after administration | 0 minute to 72 hours after administration

SECONDARY OUTCOMES:
Area under the curve of pain intensity and time in exercise (or cough) state in 0-12h, 12-24h, 12-48h and 12-72h after administration | 0 minute to 72 hours after administration
Area under the curve of pain intensity and time in resting state in 0-12h, 12-24h, 12-48h, 12-72h and 0-72h after administration | 0 minute to 72 hours after administration
Pain intensity scores in resting state and exercise (or cough) state, including within 30 minutes after anesthesia recovery and various time points after administration (6h, 8h, 12h, 18h, 24h, 30h, 36h, 48h, 72h) | recovery from anesthesia to 72 hours after administration
The duration of the first pain intensity score ≥4 points during exercise (or cough) after anesthesia recovery | 0 minute to 72 hours after administration
The duration of the first pain intensity score ≥4 points at rest after anesthesia recovery | 0 minute to 72 hours after administration
Maximum pain intensity score during exercise (or cough) within 72 hours after administration | 0 minute to 72 hours after administration
Percentage of painless (pain intensity score ≤1 at rest) subjects at planned time points | 0 minute to 72 hours after administration
Proportion of subjects who did not use remedial analgesia in 0-12h, 12-24h, 24-48h, 48-72h, 0-72h | 0 minute to 72 hours after administration
Cumulative use of remedial analgesics in 0-12h, 12-24h, 24-48h, 48-72h, 0-72h | 0 minute to 72 hours after administration
Time of first use of remedial analgesics | The time of the first pain intensity rating to 72 hours after administration
  The first time additional analgesic medication is required due to insufficient analgesic efficacy.
Subjects' analgesic satisfaction scores | 72 hours after administration
Investigators' analgesic satisfaction scores | 72 hours after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided